CLINICAL TRIAL: NCT05014139
Title: A Study of Intravesical Enfortumab Vedotin For Treatment of Patients With Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was discontinued for strategic reasons. Decision was not based on safety concerns, futility, or request from regulatory authority, ethics committee, or institutional review board or EC/IRB.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGN22E-004; EV-104 (Other: Seagen, Inc.); C5701004 (Other: Pfizer); 2023-503388-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Urinary Bladder Neoplasms; Carcinoma in Situ; Carcinoma Transitional Cell; Non-muscle Invasive Bladder Cancer; NMIBC
Keywords: Bladder Cancer; Urothelial Cancer; Enfortumab vedotin; PADCEV; Pharmacokinetics
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma in Situ; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enfortumab vedotin: Dose escalation cohort (Experimental): During the induction phase, participants will receive enfortumab vedotin once a week for 6 weeks. During the maintenance phase, participants will receive enfortumab vedotin once a month for 9 doses.
  Interventions: Drug: Enfortumab vedotin
- Enfortumab vedotin: Dose expansion cohort (Experimental): During the induction phase, participants will receive enfortumab vedotin once a week for 6 weeks. During the maintenance phase, participants will receive enfortumab vedotin once a month for 9 doses.
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Given into the bladder (intravesically)
  Other Names: PADCEV, ASG-22CE, ASG-22ME

SUMMARY:
This study will test a drug called enfortumab vedotin in participants with a type of bladder cancer called non-muscle invasive bladder cancer (NMIBC).

This study will also evaluate what the side effects are and if the drug works to treat NMIBC. A side effect is anything a drug does to your body besides treating your disease.

In this study enfortumab vedotin will be put into the bladder using a catheter. A catheter is a thin tube that can be put into your bladder.

DETAILED DESCRIPTION:
The study will be comprised of 2 parts. The first part (dose escalation) will find the highest dose of enfortumab vedotin that does not cause unacceptable side effects in participants. The second part (dose expansion) will use the dose found in the first part to test how well the drug works.

All participants will receive enfortumab vedotin. Treatment on the study will occur during the induction and maintenance phases, and participants will enter a follow-up period after completion of the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, non-muscle invasive urothelial carcinoma with carcinoma in situ (CIS) (with or without papillary disease)
* Predominant histologic component (>50 percent) must be urothelial (transitional cell) carcinoma
* Participants must have high-risk Bacillus Calmette-Guerin (BCG) - unresponsive disease, defined as (where adequate BCG therapy is defined as one of the following: 5 of 6 doses of an initial induction course + at least 2 of 3 doses maintenance therapy or 5 of 6 doses of an initial induction course + at least 2 of 6 doses of a second induction course):

  * Persistent or recurrent CIS alone or with recurrent Ta/T1 (noninvasive papillary disease/tumor invades the subepithelial connective tissue) disease within 12 months of completion of adequate BCG therapy.
  * Recurrent high-grade Ta/T1 disease within 6 months of completion of adequate BCG therapy, or
  * T1 high-grade disease at the first evaluation following an induction BCG course (at least 5 or 6 doses)
* Participant must be ineligible for or refusing a radical cystectomy
* All visible papillary Ta/T1 tumors must be completely resected within 60 days prior to enrollment.
* Eastern Cooperative Oncology Group Performance Status score of 0, 1, or 2.

Exclusion Criteria:

* Current or prior history of muscle-invasive urothelial carcinoma or metastatic disease.
* Nodal or metastatic disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) within 3 months prior to study treatment
* Concomitant upper tract urothelial carcinoma as noted on CT or MRI urogram performed within 3 months prior to study treatment
* Prior or concomitant urothelial carcinoma of the prostatic urethra within 6 months prior to study treatment
* Participants with tumor-related hydronephrosis
* Participant has received other systemic anticancer therapy including chemotherapy, biologic therapy, immunotherapy, targeted therapy, endocrine therapy, and/or investigational agent within 4 weeks or intravesical therapy within 6 weeks of first dose of study treatment
* Participant has had any prior radiation to the bladder for urothelial cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Approximately 1 year
  An AE is any untoward medical occurrence in a subject or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of laboratory abnormalities | Approximately 1 year
  To be summarized using descriptive statistics.
Incidence of dose limiting toxicities (DLTs) | Approximately 7 weeks
  To be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of enfortumab vedotin: Area under the concentration-time curve (AUC) | Approximately 1 year
  AUC will be recorded from the PK blood samples collected.
PK of enfortumab vedotin: Maximum concentration (Cmax) | Approximately 1 year
  Cmax will be recorded from the PK blood samples collected.
PK of enfortumab vedotin: Time to maximum concentration concentration (tmax) | Approximately 1 year
  Tmax will be recorded from the PK blood samples collected.
PK of enfortumab vedotin: Apparent terminal half-life (t1/2) | Approximately 1 year
  T1/2 will be recorded from the PK blood samples collected.
PK of enfortumab vedotin: Trough concentration (Ctrough) | Approximately 1 year
  Ctrough will be recorded from the PK blood samples collected.
Incidence of antitherapeutic antibodies (ATAs) to enfortumab vedotin | Approximately 1 year
  Blood samples for ATA analysis will be collected.
Complete response (CR) rate | Up to 24 months
  CR rate is defined as the proportion of subjects achieving CR.
Duration of CR | Up to 5 years
  The time from first documented CR to the first evidence of recurrence, progression, or death due to any cause.
Rate of cystectomy | Up to 5 years
  The proportion of subjects who subsequently undergo cystectomy.
Progression-free survival | Up to 5 years
  The time from start of study treatment to the first evidence of progression or death due to any cause.
Cystectomy-free survival | Up to 5 years
  The time from start of study treatment to cystectomy or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (21):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - UCLA Department of Medicine - Hematology & Oncology, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California at San Francisco, San Francisco, California
  - Stanford Health Care, Stanford, California
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Markey Cancer Center / University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Erlanger Oncology and Hematology, Chattanooga, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Fred Hutchinson Cancer Center / Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
- Site CA11001, Toronto, Ontario, Canada
- France (3):
  - Site FR33002, Lyon
  - Site FR33001, Paris
  - Site FR33003, Rennes
- Germany (2):
  - Site DE49001, Göttingen
  - Site DE49002, Tübingen
- Spain (4):
  - Site ES34001, Barcelona
  - Site ES34004, Barcelona
  - Site ES34003, Barcelona
  - Site ES34002, Madrid
- Site UK44002, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No